CLINICAL TRIAL: NCT04240275
Title: Reliability of a Body-worn Sensor System for Analysis of Spatiotemporal Gait Parameters in Children With CP
Brief Title: Reliability of a Body-worn Sensor System for Gait Analysis in Children With CP
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Gokhan Yazici, Principal Investigator, Gazi University
Other Study IDs: 12355
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Cerebral Palsy, Spastic; Gait Disorders, Neurologic
Keywords: Cerebral Palsy; Gait Assessment; G-Walk; Reliability
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic | interventions — Gait Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with Cerebral Palsy: Children diagnosed with Spastic Cerebral Palsy (Unilateral or Bilateral) among the age range of 5-15 who can walk independently
  Interventions: Device: Reliability of the G-Walk device in children with Cerebral Palsy

INTERVENTIONS:
Device: Reliability of the G-Walk device in children with Cerebral Palsy — The purpose of this study was to confirm the test-retest reliability of a commercially available body-worn sensor-G-Walk® sensor system-for spatiotemporal gait parameters in children with CP.
  The children will be assessed with the G-Walk on two separate occasions.For the reliability analysis, the second measurement tests will be repeated 3 days after the first assessment.
  The device is placed on an elastic belt and worn on the waist of the person being evaluated, with the center of the device at the fifth lumbar vertebrae. To ensure correct placement of the device, the L4-L5 intervertebral space will be palpated via the posterior superior iliac spines (SIPS).
  After the accelerometer is placed, the children are asked to walk calmly at normal speed, on a 10 m track, whose boundaries will be determined with colored lines and to return to the starting position.
  Other Names: Gait Analysis

SUMMARY:
Cerebral palsy (CP) is caused by a non-progressive injury in the developing brain, which leads to problems in functional mobility, posture, neuro musculoskeletal functions and gait. Around 75% of children with CP are ambulatory however they have gait problems such as excessive knee flexion, stiff knee, crouch gait or equinus which affects the quality of gait. When constructing an effective treatment plan in children with CP, a comprehensive assessment should be performed. One of the most essential assessments is gait analysis. Gait analysis is used in the quantitative assessment of gait disturbances providing functional diagnosis, assessment for treatment, planning, and monitoring of progress.

Gait analysis aims to determine the factors leading to gait disturbances. To reach this aim, a large amount of quantitative data concerning the gait characteristics of a patient is analyzed. The assessment of these data can be performed via standardized clinical videos, recorded with numerical video cameras used in conjunction with optical 3D systems. The purpose of this study was to confirm the test-retest reliability of a commercially available body-worn sensor- G-Walk® sensor system-for spatiotemporal gait parameters in children with CP.

DETAILED DESCRIPTION:
The G-Walk determines spatiotemporal parameters as well as pelvic rotations during gait and allows objective and precise analysis of movements with its wearable inertial sensor. It also enables 3D kinematic analysis of the pelvis, providing a functional analysis of disorders in gait caused by neuromuscular diseases The device is placed on an elastic belt and worn on the waist of the person being evaluated, with the center of the device at the fifth lumbar vertebrae. To ensure correct placement of the device, the L4-L5 intervertebral space was palpated via the posterior superior iliac spines (SIPS).

After the accelerometer was placed, the children were asked to walk calmly at normal speed, on a 10 m track, whose boundaries were determined with colored lines and to return to the starting position.

The values and gait characteristics of acceleration in the anteroposterior (AP) and mediolateral (ML) axes were transferred to the computer software program.

The tilt of the pelvis in the sagittal plane in the flexion-extension direction, the oblique displacement in the coronal plane, the angles of the rotation of movement in the transverse plane and the symmetry values of the right and left sides are obtained. While the symmetry index ranges from 0 to 100, a value closer to 100 indicates that the gait is more symmetrical

ELIGIBILITY:
Inclusion Criteria:

* Accepting to participate in the study,
* Being between 5-15 years old,
* Having a diagnosis of Spastic Cerebral Palsy,
* Being level I-II according to GMFCS

Exclusion Criteria:

* Having limited cooperation which prevents participation in the study,
* Refusing to participate in the study,
* Having an orthopedic disorder or systemic illness which prevents movement in the lower extremities,
* Having a Botulinum toxin application in the last 3 month

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with Spastic Cerebral Palsy who have involvement on one or two sides of the body, who can walk independently.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Gait Symmetry | Reliability of the G-Walk in 3 days
  Gait parameters will be assessed via the G-Walk on two separate occasions. The G-Walk is a device that is worn on the waist via an elastic belt. The G-Walk is built with a triaxial accelerometer 16 bit/axes with multiple sensitivity, a triaxial magnetometer 13 bit and a triaxial gyroscope 16 bit/axes with multiple sensitivity. This hardware is capable of acquiring and transmitting data to a computer through a Bluetooth connection and at the end of each analysis an automatic report containing the gait assessment results is ready to be analyzed.
  Gait symmetry values of the right and left sides are obtained within this report. While the symmetry index ranges from 0 to 100, a value closer to 100 indicates that the gait is more symmetrical.
Gait Speed | Reliability of the G-Walk in 3 days
  Gait parameters will be assessed via the G-Walk on two separate occasions. The G-Walk is a device that is worn on the waist via an elastic belt. The G-Walk is built with a triaxial accelerometer 16 bit/axes with multiple sensitivity, a triaxial magnetometer 13 bit and a triaxial gyroscope 16 bit/axes with multiple sensitivity. This hardware is capable of acquiring and transmitting data to a computer through a Bluetooth connection and at the end of each analysis an automatic report containing the gait assessment results is ready to be analyzed.
  For each subject, mean gait speed will be calculated from 10 consecutive steps in the gait cycles.
Spatiotemporal gait parameters | Reliability of the G-Walk in 3 days
  Gait parameters will be assessed via the G-Walk on two separate occasions. The G-Walk is a device that is worn on the waist via an elastic belt. The G-Walk is built with a triaxial accelerometer 16 bit/axes with multiple sensitivity, a triaxial magnetometer 13 bit and a triaxial gyroscope 16 bit/axes with multiple sensitivity. This hardware is capable of acquiring and transmitting data to a computer through a Bluetooth connection and at the end of each analysis an automatic report containing the gait assessment results is ready to be analyzed.
  The device provides the data for the following spatiotemporal gait parameters in one single report; Cadence Stance Phase (%of gait) Swing Phase (%of gait) Stride Length (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Gokhan Yazici, Pt. PhD, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data will not be available to other researchers.

REFERENCES:
- [Background] De Ridder R, Lebleu J, Willems T, De Blaiser C, Detrembleur C, Roosen P. Concurrent Validity of a Commercial Wireless Trunk Triaxial Accelerometer System for Gait Analysis. J Sport Rehabil. 2019 Aug 1;28(6):jsr.2018-0295. doi: 10.1123/jsr.2018-0295. PMID 30747572
- [Background] Kleiner AFR, Pacifici I, Vagnini A, Camerota F, Celletti C, Stocchi F, De Pandis MF, Galli M. Timed Up and Go evaluation with wearable devices: Validation in Parkinson's disease. J Bodyw Mov Ther. 2018 Apr;22(2):390-395. doi: 10.1016/j.jbmt.2017.07.006. Epub 2017 Jul 25. PMID 29861240
- [Background] Armand S, Decoulon G, Bonnefoy-Mazure A. Gait analysis in children with cerebral palsy. EFORT Open Rev. 2016 Dec 22;1(12):448-460. doi: 10.1302/2058-5241.1.000052. eCollection 2016 Dec. PMID 28698802